CLINICAL TRIAL: NCT03908606
Title: Prognostic Value of Serum Hs-CRP in Periodontitis Patients With or Without Type 2 Diabetes Following Non-surgical Periodontal Therapy
Brief Title: Serum Hs-CRP in Periodontitis Patients With or Without Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Gihane Gharib Madkour, Associate professor, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1281976
Record Dates: First submitted 2019-04-06; First posted 2019-04-09 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Periodontal Disease; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Periodontal Diseases; Diabetes Mellitus, Type 2 | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Periodontitis patients with diabetes type 2 (Experimental): scaling and root planing was administered to all patients. Serum samples were collected before and after treatment to assess hs-CRP levels. Glycated hemoglobin was measured before and after treatment
  Interventions: Procedure: Scaling and root planing
- Periodontitis patients (Experimental): scaling and root planing will be done to periodontitis patients. Serum samples were collected before and after treatment to assess hs-CRP levels.
  Interventions: Procedure: Scaling and root planing
- Healthy control group (No Intervention): We measured serum levels of hs-CRP in all healthy control subjects

INTERVENTIONS:
Procedure: Scaling and root planing — Supra and subgingival scaling and root planing.
  Arms: Periodontitis patients; Periodontitis patients with diabetes type 2

SUMMARY:
the aim of this study was to assess serum levels of high sensitivity c reactive protein in periodontitis patients with and without type 2 diabetes in a trial to analyze its prognostic effect following non-surgical periodontal therapy.

DETAILED DESCRIPTION:
Periodontitis and diabetes are chronic disorders with a two-way correlation as they can both stimulate an inflammatory response with subsequent formation of inflammatory mediators and cytokines. C reactive protein is an inflammatory plasma marker having a role in the systemic reaction to inflammation. thus, our aim in the current study was to evaluate serum levels of high sensitivity c reactive protein in periodontitis patients with and without type 2 diabetes in a trial to analyze its prognostic effect following non-surgical periodontal therapy. A total of 60 patients were enrolled in this study. ELISA was used for determination of hs- CRP. Non- surgical periodontal therapy was carried out for all periodontitis patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetic patients type 2
2. Periodontitis patients

Exclusion Criteria:

1. Smokers
2. Pregnant females

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-01-02 (Actual)

PRIMARY OUTCOMES:
clinical attachment level | 3 months
  gain in clinical attachment level

CONTACTS AND LOCATIONS:
Overall Officials: Gihane Madkour, Prof, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No